CLINICAL TRIAL: NCT00025077
Title: Treatment Of Recurrent Central Nervous System Primitive Neuroectodermal Tumors (PNETs) In Children And Adolescents A Strategy Including The Use Of High Dose Thiotepa And High Dose Carboplatin
Brief Title: Combination Chemotherapy, Surgery or Radiation Therapy, and Peripheral Stem Cell Transplant in Treating Patients With Recurrent Medulloblastoma or Primitive Neuroectodermal and Pineal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CCLG-CNS-2000-01; CDR0000068910 (Registry Identifier: PDQ (Physician Data Query)); EU-20105
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2007-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood medulloblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Medulloblastoma | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Thiotepa; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: thiotepa
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug before surgery or radiation therapy may shrink the tumor so that it can be removed during surgery or radiation therapy. Peripheral stem cell transplant may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy and allow doctors to give higher doses of chemotherapy.

PURPOSE: This phase II trial is studying how well combination chemotherapy followed by surgery or radiation therapy and peripheral stem cell transplant work in treating patients with recurrent medulloblastoma or primitive neuroectodermal and pineal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of cyclophosphamide and surgical resection or radiotherapy followed by thiotepa, carboplatin, and autologous peripheral blood stem cell rescue in patients with recurrent medulloblastoma or supratentorial neuroectodermal and pineal tumors.
* Determine the acute and chronic toxicity of this regimen in these patients.
* Determine progression-free and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Cytoreductive Phase: Patients receive cyclophosphamide IV over 1 hour on days 1 and 2 and filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 7 and continuing until blood counts recover. Treatment repeats after discontinuation of G-CSF for 2-4 courses. Peripheral blood stem cells (PBSC) are harvested after each course of cyclophosphamide. Patients undergo surgical resection or radiotherapy after the completion of chemotherapy. Patients achieving complete response proceed to myeloablative therapy.
* Myeloablative Phase: Patients receive thiotepa IV over 3 hours on days 1-3. Autologous PBSC are reinfused on day 5 and patients receive G-CSF SC once daily beginning on day 10 and continuing until blood counts recover. Beginning 2 days after the completion of G-CSF, patients receive carboplatin IV over 1 hour on days 1-3. Autologous PBSC are reinfused on day 5 and patients receive G-CSF SC once daily beginning on day 10 and continuing until blood counts recover.

Patients are followed at 1, 3, 6, and 12 months.

PROJECTED ACCRUAL: Approximately 50 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent medulloblastoma or supratentorial primitive neuroectodermal and pineal tumor

  * Nodular/desmoplastic medulloblastoma
  * Medullomyoblastoma
  * Melanotic medulloblastoma
  * Ependymoblastoma
  * Pinealoblastoma
* Received prior craniospinal radiotherapy OR
* Relapse in site of prior localized radiotherapy (e.g., relapse after "baby brain" protocol)

PATIENT CHARACTERISTICS:

Age:

* Under 21

Performance status:

* Lansky 40-100% for ages 1-16 years
* Karnofsky 40-100% for ages over 16 years

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than upper limit of normal (ULN)
* AST less than 2 times ULN

Renal:

* Glomerular filtration rate at least 60 mL/min

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2000-01; Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Event-free survival

SECONDARY OUTCOMES:
Toxic death rate

CONTACTS AND LOCATIONS:
Overall Officials: Barry Pizer, MD, Study Chair — Royal Liverpool Children's Hospital, Alder Hey
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - University College of London Hospitals, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton University Hospital NHS Trust, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland